CLINICAL TRIAL: NCT06218563
Title: Vibration-induced Movement Illusion Causes Cerebral Haemodynamic Changes: A fNIRS Study.
Brief Title: Study of Cerebral Activation by fNIRS During Vibration-induced Illusion of Movement in Healthy and Stroke Participants.
Acronym: VIBRANIRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHRO-2023-05
Record Dates: First submitted 2024-01-12; First posted 2024-01-23 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Healthy; Stroke, Acute
Keywords: Vibration; Illusion of movement; Functional Near Infrared Spectroscopy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: The protocol consists of 4 or 2 different conditions (repeated 2 times) of vibration-induced illusion of movement in healthy and stroke participants respectively, resulting in 8 or 4 vibration blocks with 3 vibrations per block.
  Conditions order is pseudorandomized, participants can start by the left or the right arm with eyes opened or closed. When starting with either the left or right arm, all conditions are completed before moving on to the other arm (for healthy participants). In total, the number of participants starting with right or left vibration should be the same.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- vibration-induced illusion of movement (Experimental): The protocol consists of 4 or 2 different conditions (repeated 2 times) of vibration-induced illusion of movement in healthy and stroke participants respectively, resulting in 8 or 4 vibration blocks with 3 vibrations per block:
  Healthy participants, 2 times each (24 vibrations):
  * Right arm, eyes opened (no-illusion condition; RO)
  * Right arm, eyes closed (illusion condition; RC)
  * Left arm, eyes opened (no-illusion condition; LO)
  * Left arm, eyes closed (illusion condition; LC)
  Stroke participants, 2 times each (12 vibrations):
  * Deficient side, eyes opened (no-illusion condition; DO)
  * Deficient side, eyes closed (illusion condition; DC)
  Interventions: Other: vibration-induced illusion of movement

INTERVENTIONS:
Other: vibration-induced illusion of movement — Conditions order is pseudorandomized, participants can start by the left or the right arm with eyes opened or closed. When starting with either the left or right arm, all conditions are completed before moving on to the other arm (for healthy participants). In total, the number of participants starting with right or left vibration should be the same.

SUMMARY:
The purpose of this study is to investigate the cerebral activation of healthy and stroke participants in 4 or 2 different conditions (repeated 2 times) of vibration-induced illusion of movement respectively, resulting in 8 or 4 vibration blocks with 3 vibrations per block. The frequency of the vibration being 80 Hz.

Healthy participants:

* Right arm, eyes opened
* Right arm, eyes closed
* Left arm, eyes opened
* Left arm, eyes closed

Stroke participants:

* Deficient side, eyes opened
* Deficient side, eyes closed

The aim is to compare the subjective sensation of movement score and cerebral activations of healthy/stroke participants depending on the condition.

DETAILED DESCRIPTION:
Perceived sensations of limb and movements (kinesthesia) allow us to situate ourselves without visual feedback and not dedicate all of our attention to everyday tasks such as walking or taking and holding an object. These perceived conscious sensations come from receptors called proprioceptors which are located in the skin, joints and muscles. When a limb is moving and a muscle is stretched, the main sensation of limb stretching comes from the stimulation of a proprioceptor called the muscle spindle, more specifically from its primary ending called the 1a fibber. Artificially, 1a fibbers can be (optimally) stimulated by vibration of the muscle around 80 Hz. When stimulating 1a fibbers of the triceps, a signal of stretching is produced and an illusion of flexion can be felt as long as their no other contrary feedback involved such as vibration of the antagonist muscle or visual feedback of the immobile limb as it provides a more reliable information to the brain. As of now, neural correlates to muscle spindle vibration and illusion of movement have not been fully characterize in healthy participants and are not known in stroke participants.

To investigate the effect of vibration-induced illusion of movement on cerebral activations in healthy and stroke participants, the investigators propose to use an innovative tool of neuroimaging, the functional near infrared spectroscopy (fNIRS).

fNIRS allows to investigate cortical cerebral activations by measuring cerebral haemodynamic variations. Indeed, just like fMRI, it relies on the haemodynamic response function (HRF) caused by neurovascular coupling. Its portability and non-invasiveness make it a great tool to study brain activations in a more ecological environment (in a standing or sitting position for example).

This research aims to study and compare the subjective sensation of movement and the cortical cerebral areas involved in muscle spindle vibration and illusion of movement in healthy and stroke participants.

The protocol consists of 4 or 2 different conditions (repeated 2 times) of vibration-induced illusion of movement in healthy and stroke participants respectively, resulting in 8 or 4 vibration blocks with 3 vibrations per block:

Healthy participants, 2 times each (24 vibrations):

* Right arm, eyes opened (no-illusion condition; RO)
* Right arm, eyes closed (illusion condition; RC)
* Left arm, eyes opened (no-illusion condition; LO)
* Left arm, eyes closed (illusion condition; LC)

Stroke participants, 2 times each (12 vibrations):

* Deficient side, eyes opened (no-illusion condition; DO)
* Deficient side, eyes closed (illusion condition; DC)

Conditions order is pseudorandomized, participants can start by the left or the right arm with eyes opened or closed. When starting with either the left or right arm, all conditions are completed before moving on to the other arm (for healthy participants). In total, the number of participants starting with right or left vibration should be the same.

The fNIRS devices that will be used are the Brite MKII and Brite MKIII (Artinis Medical system, Netherlands).

The vibration tool that will be used is a vibrator from VibraMoov. The subjective sensation of movement will be analyzed using the Standardized Kinesthetic Illusion Procedure (SKIP) scale. Participants will have to report their sensation of movement after each condition (3 vibrations block) from 0 to 3, 0 being no sensation of movement and 3 being a clear and precise sensation of movement. Participants will also have to describe the direction of movement, a score of 1 will be attributed if the movement described correspond to the one expected and a score of 0 will be attributed for every other movements.

ELIGIBILITY:
Inclusion Criteria:

* 18-85 years old
* Able to sign a consent form
* Sufficient command of the French language to understand instructions
* Affiliated to a social security scheme

Healthy participants:

* Right handed
* No neurological disease or motor deficit

Stroke participants:

* Stroke volunteers in acute phase (before day 14 post-stroke)
* Not aphasic
* Able to maintain sitting position without difficulty
* Deficit moteur
* Able to sign a consent form

Exclusion Criteria:

* Person under tutorship or curatorship
* Known allergy to of the fNIRS cap components: neoprene
* No vibrations feeling on the deficient side
* Vigilance-modifying drugs (high-dose psychotropics, antispastic drugs)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2025-06-25 (Actual); Study Completion 2025-06-25 (Actual)

PRIMARY OUTCOMES:
Mean change in the concentration of oxyhemoglobin during the task | Day 0
  The HbO2 signals are considered as indicators of the hemodynamic response.
Mean change in the concentration of deoxyhemoglobin during the task | Day 0
  The HbR signals are considered as indicators of the hemodynamic response.

SECONDARY OUTCOMES:
SKIP scale | Day 0
  The subjective sensation of movement will be analyzed using the Standardized Kinesthetic Illusion Procedure (SKIP) scale. Participants will have to report their sensation of movement after each condition (3 vibrations block) from 0 to 3, 0 being no sensation of movement and 3 being a clear and precise sensation of movement. Participants will also have to describe the direction of movement, a score of 1 will be attributed if the movement described correspond to the one expected and a score of 0 will be attributed for every other movements.

CONTACTS AND LOCATIONS:
Overall Officials: Canan OZSANCAK, Dr, Principal Investigator — CHU d'Orléans
Locations (1):
- CHU d'ORLEANS, Orléans, France

REFERENCES:
- [Background] Adamo DE, Scotland S, Martin BJ. Upper limb kinesthetic asymmetries: gender and handedness effects. Neurosci Lett. 2012 May 16;516(2):188-92. doi: 10.1016/j.neulet.2012.03.077. Epub 2012 Apr 3. PMID 22490887
- [Background] Chancel M, Landelle C, Blanchard C, Felician O, Guerraz M, Kavounoudias A. Hand movement illusions show changes in sensory reliance and preservation of multisensory integration with age for kinaesthesia. Neuropsychologia. 2018 Oct;119:45-58. doi: 10.1016/j.neuropsychologia.2018.07.027. Epub 2018 Jul 29. PMID 30063911
- [Background] Collins DF, Refshauge KM, Todd G, Gandevia SC. Cutaneous receptors contribute to kinesthesia at the index finger, elbow, and knee. J Neurophysiol. 2005 Sep;94(3):1699-706. doi: 10.1152/jn.00191.2005. Epub 2005 May 25. PMID 15917323
- [Background] Desmurget M, Reilly KT, Richard N, Szathmari A, Mottolese C, Sirigu A. Movement intention after parietal cortex stimulation in humans. Science. 2009 May 8;324(5928):811-3. doi: 10.1126/science.1169896. PMID 19423830
- [Background] Gilhodes JC, Roll JP, Tardy-Gervet MF. Perceptual and motor effects of agonist-antagonist muscle vibration in man. Exp Brain Res. 1986;61(2):395-402. doi: 10.1007/BF00239528. PMID 3948946
- [Background] Guerraz M, Provost S, Narison R, Brugnon A, Virolle S, Bresciani JP. Integration of visual and proprioceptive afferents in kinesthesia. Neuroscience. 2012 Oct 25;223:258-68. doi: 10.1016/j.neuroscience.2012.07.059. Epub 2012 Aug 3. PMID 22864182
- [Background] Hagura N, Takei T, Hirose S, Aramaki Y, Matsumura M, Sadato N, Naito E. Activity in the posterior parietal cortex mediates visual dominance over kinesthesia. J Neurosci. 2007 Jun 27;27(26):7047-53. doi: 10.1523/JNEUROSCI.0970-07.2007. PMID 17596454
- [Background] Imai R, Hayashida K, Nakano H, Morioka S. Brain Activity Associated with the Illusion of Motion Evoked by Different Vibration Stimulation Devices: An fNIRS Study. J Phys Ther Sci. 2014 Jul;26(7):1115-9. doi: 10.1589/jpts.26.1115. Epub 2014 Jul 30. PMID 25140108
- [Background] Kodama T, Nakano H, Ohsugi H, Murata S. Effects of vibratory stimulation-induced kinesthetic illusions on the neural activities of patients with stroke. J Phys Ther Sci. 2016 Jan;28(2):419-25. doi: 10.1589/jpts.28.419. Epub 2016 Feb 29. PMID 27065525
- [Background] Proske U, Gandevia SC. The proprioceptive senses: their roles in signaling body shape, body position and movement, and muscle force. Physiol Rev. 2012 Oct;92(4):1651-97. doi: 10.1152/physrev.00048.2011. PMID 23073629
- [Background] Romaiguere P, Anton JL, Roth M, Casini L, Roll JP. Motor and parietal cortical areas both underlie kinaesthesia. Brain Res Cogn Brain Res. 2003 Mar;16(1):74-82. doi: 10.1016/s0926-6410(02)00221-5. PMID 12589891
- [Background] Skinner HB, Barrack RL, Cook SD. Age-related decline in proprioception. Clin Orthop Relat Res. 1984 Apr;(184):208-11. PMID 6705349
- [Background] Tidoni E, Fusco G, Leonardis D, Frisoli A, Bergamasco M, Aglioti SM. Illusory movements induced by tendon vibration in right- and left-handed people. Exp Brain Res. 2015 Feb;233(2):375-83. doi: 10.1007/s00221-014-4121-8. Epub 2014 Oct 8. PMID 25294499
- [Derived] Leger B, Auzou P, Fourdrinoy E, Sarrazin M, Celot S, Gay C, de Dieuleveult B, Cohen C, Perrey S, Ozsancak C. Vibration-induced illusion of movement is hindered by acute stroke but mostly by aging: a cross-sectional study. Aging Clin Exp Res. 2025 Dec 1;38(1):20. doi: 10.1007/s40520-025-03247-6. PMID 41324779